CLINICAL TRIAL: NCT06595927
Title: Comparison and Correlation of Clinical Signs With Changes in the Activity of the Cervical Muscles Evaluated by Muscle Functional Magnetic Resonance Imaging During the Cervical Cervical Extensor Endurance Test
Brief Title: Clinical Signs and Changes in Cervical Muscles Activity Evaluated by Magnetic Resonance Imaging During an Endurance Test
Acronym: CEET/IRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Colman (Other)
Collaborators: University of Liege (Other)
Responsible Party: Sponsor-Investigator, David Colman, PhD student, Principal Investigator, University of Liege
Organization: University of Liege (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: B7072021000028
Record Dates: First submitted 2022-08-23; First posted 2024-09-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain; Motor Activity
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Recruitment Detection, Audiologic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with chronic neck pain (Experimental): Both groups will receive the same experimental procedure, divided in 2 parts.
  Part 1: a first cervical MRI is done, followed by a cervical extensor endurance test during 3 minutes and the second cervical MRI.
  Part 2 : several clinical tests will be done:
  * tandem stand balance test (eyes closed, firm ground)
  * cranio-cervical flexion test
  * head lift test
  * cervical joint position error sense test in 4 directions
  Interventions: Diagnostic Test: Cervical extensor endurance test
- Participants free of neck pain (Active Comparator): the same experimental procedure than the other group
  Interventions: Diagnostic Test: Cervical extensor endurance test

INTERVENTIONS:
Diagnostic Test: Cervical extensor endurance test — Monitoring the clinical parameters of head and neck immobility during the cervical extensor endurance test to correlate them with muscular activity by MRI and other cervical clinical tests
  Other Names: cervical flexor muscles motor control tests; balance test; cervical proprioception test

SUMMARY:
The aim of this present study is to compare the radio-clinic correlation between the ability to hold the head and neck (by inertial sensor) and the changes in neck muscles activity (by functional magnetic resonance imaging) during the cervical extensor endurance test between an asymptomatic population and one suffering from chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Neck Disability Index score > 8/50 for the symptomatic group OR < 4/50 for the asymptomatic group
* numerical rating scale < 7/10 for the symptomatic group
* suffering from idiopathic or traumatic chronic neck pain for the neck pain group OR being free of neck pain which required therapeutic, medical or medicinal treatment in the last 12 months.

Exclusion Criteria:

* fibromyalgia, cervical radiculopathy, previous cervical surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Change of Cervical muscles metabolism by the transverse relaxation time (T2) values in milliseconds | At baseline and after the endurance test, to assess the change of T2 values
  The MRI, after identifying the region of interest for each muscle, will be used to calculate a transverse relaxation time (T2) value (in milliseconds) for each muscle at two assessment points: before and after the cervical extensor endurance test. The aim is to evaluate the changes in T2 values induced by each muscle's contribution during the endurance test. Each MRI scan will last 11 minutes.
Head and neck movements in degrees or millimetres during the cervical extensor endurance test. | At baseline (just after the first MRI)
  The inertial sensor will monitor the head and neck movements during the entire duration of the Cervical Extensor Endurance Test, in the three planes of space for cervical movements and for cranio-cervical flexion/extension movement.
  The maximal duration of 3 minutes of the cervical extensor endurance test

SECONDARY OUTCOMES:
Tandem stand balance test in seconds | During the 7 days following the MRI
  The participant must stand with both feet bare on the floor, aligning them so that the big toe of the back foot is in contact with the heel of the front foot, knees straight and eyes closed.
  The aim is to hold this position for 30 seconds without changing feet or reopening the eyes.a stopwatch is used to evaluate this test, during 30 seconds maximum.
Cervical joint position sense error test in millimetres | During the 7 days following the MRI
  The participant sits on a chair with a backrest, a helmet with a laser pointing forward is placed on his head.
  A target is placed in front of him/her, against a wall 90 cm from the participant's forehead, so that the laser points to the centre of the target when the participant is in a comfortable neutral position.
  The participant's ability to reposition himself in this neutral position is assessed by asking him to perform 6 successive movements of left, right rotation, flexion and then extension, before returning to the centre of the target, as close as possible to the starting position. These movements will all be performed with the eyes closed.
  The offset between the return position and the starting position will be assessed by measuring the distance in millimetres from the centre of the target to the return position of the laser.
  The next movement will only be performed after a return to the neutral position, performed passively by the experimenter.
Head lift test in seconds | During the 7 days following the MRI
  The participant lies on his or her back with arms at his or her side and knees bent so that the feet are flat on the examination table, without a pillow.
  The examiner places a two-finger thickness between the participant's external occipital protuberance and the table.
  The participant is asked to perform maximum craniocervical flexion combined with cervical and cervicothoracic global flexion in order to touch the examiner's fingers under the head.
  He must maintain the position as long as possible, without rising or falling and without losing the cranio-cervical flexion position. The test is therefore measured in seconds with a stopwatch. The longer the duration, the better.
Cranio-cervical flexion test in mmHg | During the 7 days following the MRI
  The participant lies on his back with arms at his sides The test tool, a Stabilizer, is folded in 3 layers and placed just below the sub-occipital ridges and inflated so that the needle reads 20 mmHg in the starting position The participant is asked to actively perform a slow, measured craniocervical flexion so that he can reach the following graduations successively over a period of 2 to 3 seconds: 22 mmHg, 24 mmHg, 26 mmHg, 28 mmHg and 30 mmHg, starting each trial at 20 mmHg. The higher the level reached correctly, the better.
  The test stops when the participant: fails to reach/hold the required level for 2 - 3 seconds, performs a retraction movement to reach the required level, performs a thoracic extension to reach the required level or uses superficial cervical muscle activity (sternocleidomastoid, anterior scalene) to reach the required level. In this case, the last stop (in mmHg) reached correctly is taken as an indicator of the level of performance for this test.
Endurance in cranio-cervical flexion test (in percent) | During the 7 days following the MRI
  The participant lies on his or her back with arms at his sides. The test tool, the Stabilizer, and placed just below the sub-occipital ridges and inflated so that the needle reads 20 mmHg in the starting position The participant is asked to actively perform a slow craniocervical flexion in order to realize 10 repetitions of 10 seconds each, at the following pressure levels: 22, 24, 26, 28 and 30 mmHg The higher the level reached correctly, the better. The test stops when the participant: fails to reach/hold the required pressure level for 10 seconds, performs a retraction movement/ thoracic extension/ uses superficial cervical muscle (sternocleidomastoid, anterior scalene) activity to reach the required pressure level. In this case, the number of repetitions correctly performed at the last level reached are used to assess the performance as follow: each successful repetition has a value of 2%, reaching 100% at the 10th repetition performed at 30 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Marc MV Vanderthommen, Professor, Study Chair — University of Liege
Locations (1):
- University Hospital of Liege, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cagnie B, O'Leary S, Elliott J, Peeters I, Parlevliet T, Danneels L. Pain-induced changes in the activity of the cervical extensor muscles evaluated by muscle functional magnetic resonance imaging. Clin J Pain. 2011 Jun;27(5):392-7. doi: 10.1097/AJP.0b013e31820e11a2. PMID 21415716